CLINICAL TRIAL: NCT02352207
Title: Prospective Identification of Predictors of Neonatal Respiratory Distress for Newborns With Prenatally Diagnosed Congenital Lung Malformations : A Population-based, Nationally Representative Study
Brief Title: Risk Factors of Neonatal Respiratory Distress for Newborns With Prenatally Diagnosed Congenital Lung Malformations
Acronym: MALFPULM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI13005
Record Dates: First submitted 2015-01-05; First posted 2015-02-02 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Foetus With Congenital Pulmonary Malformation
Keywords: Neonatal respiratory distress; prenatal lung malformation; KRAS mutation; pregnant woman
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A portion of tissue malformation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- identification of a pulmonary malformation in the fetus: pregnant women referred to a prenatal Center, because of the identification of a pulmonary malformation in the fetus
  Interventions: Other: identification of a pulmonary malformation in the fetus

INTERVENTIONS:
Other: identification of a pulmonary malformation in the fetus

SUMMARY:
This research focuses on lung malformations detected in fetuses during prenatal ultrasound exams. Pathogenic mechanisms of these rare malformations are poorly understood. Improved knowledge is needed, to give families better information, and to better standardize treatment decisions The main goal is to better predict neonatal complications associated with these malformations, by identifying key predictive markers during the fetal period.

To achieve this objective, it is planned to include 400 pregnant women with prenatal diagnosis of pulmonary malformation in 45 health centers in France. This is the largest study on this topic at the international level.

DETAILED DESCRIPTION:
The main objective of the study is to develop a prognostic model for estimating the risk of neonatal respiratory distress in children with prenatally diagnosed congenital pulmonary malformation.

The study will be offered to all pregnant women referred to a Center for Prenatal Diagnosis (CPD), due to the identification of a congenital lung malformations in the fetus. This study does not induce any changes in clinical and therapeutic monitoring proposed by the team in charge of the mother. At inclusion, and at each prenatal evaluation, prenatal parameters are entered in an e-CRF. In an effort to minimize any potential intra- and interoperator variability in malformation measurements over time, this study includes a standardized and centralized evaluation of ultrasound and MRI (if available) acquisitions of volume measurements. When the place of delivery is determined, a contact is made before birth with the teams (maternity, neonatology, intensive care unit), so that neonatal data are also collected prospectively. A phone call to the family is planned for the end of the first postnatal month, to identify any respiratory event that would have occurred between returning home after childbirth and the first month.

The routine follow-up of these children is then ensured in accordance with current national recommendations, in conjunction with the reference centers for rare respiratory diseases in children (28 university hospitals, spread across all regions of France). A telephone survey every 6 months with the referring physician in this specialized center or, alternatively, with the family, will collect clinical outcome until the age of 2 years. If a surgical intervention is planned within this interval, consent to collect part of the surgical specimen for research purposes will be solicited. This tissue will be immediately frozen at -80 ° C, to allow laser microdissection and DNA extraction from epithelial cells lining the malformation (Inserm U955). Frozen tissue will be conserved at the biobank of Necker-Enfants Malades.

ELIGIBILITY:
Inclusion Criteria:

* Prenatal identification of a congenital pulmonary malformation (hyperechoic and/or cystic pulmonary lesion)
* consent of the mother for participation to the study

Exclusion Criteria:

- Absence of consent for participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women referred to a Center of Prenatal Diagnosis, because of the identification of a pulmonary malformation in the fetus
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Respiratory distress | At Birth of the child
  Respiratory distress at birth is defined by a breathing frequency > 60/min, or by the presence of chest retraction signs (Silverman score greater than or equal to 2). At least one of these signs must be persistent at 15' of life

SECONDARY OUTCOMES:
Necessity of antenatal treatment | At Birth of the child
  Thoracic drainage, amniotic drainage, corticosteroids
Therapeutic abortion - fetal death | At Birth of the child
Severe respiratory distress | At Birth of the child
  Severe respiratory distress at birth will be defined by the presence of at least one of the following parameters: persistent need at 15' of supplemental oxygen; Persistent need at 15' for a ventilatory support (non-invasive or invasive); neonatal death
Identification of KRAS mutation | 2 years
  PCR analysis of known K-RAS mutations in codons 12 and 13
Level in delta Forskoline/IBMX Short Circuit Current (µA/cm2) | 2 years
  CFTR activity evaluation
CFTR gene expression | 2 years
  quantitative PCR
CFTR protein expression | 2 years
  immunohistochemistry
Basal short circuit current : Isc Basal | 2 years
Effects of other potentiators on CFTR activity : ΔGenistein, ΔVX-770 | 2 years
Inhibition of CFTR (inh-172) : ΔInh-172 | 2 years
Response to ENaC inhibitors : ΔAmiloride, Δbenzamil | 2 years
Activation of Calcium Dependant Channels : ΔUTP | 2 years
Inhibition of SLC26A9 : ΔGlyH-101 | 2 years
Response to inhibitors of basolateral K+ secretion : ΔBarium ; ΔChromanol | 2 years
Secretion of HCO3- in response to forskoline : Δ HCO3- primary culture | 2 years
Gene expression of other channels : ENaC, SLC26A9, CaCC, KVLQT1 and KCa3.1 | 2 years
  quantitative PCR
Protein expression of other channels : ENaC, SLC26A9, CaCC, KVLQT1 and KCa3.1 | 2 years
  immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SALOMON, MD, PhD, Study Director — Hospital Necker - Enfants Malades
Locations (1):
- Hôpital Necker - Enfants Malades, Paris, France

REFERENCES:
- [Result] Delacourt C, Bertille N, Salomon LJ, Rahshenas M, Benachi A, Bonnard A, Choupeaux L, Fouquet V, Goua V, Hameury F, Hervieux E, Jouannic JM, Khen-Dunlop N, Le Bouar G, Massardier J, Roditis L, Rosenblatt J, Sartor A, Thong-Vanh C, Lelong N, Khoshnood B; , for the MALFPULM study group; members of the MALFPULM study group:. Predicting the risk of respiratory distress in newborns with congenital pulmonary malformations. Eur Respir J. 2022 Feb 3;59(2):2100949. doi: 10.1183/13993003.00949-2021. Print 2022 Feb. PMID 34266941
- [Result] Delacourt C, Bertille N, Salomon LJ, Benachi A, Henry E, Massardier J, Mottet N, Rosenblatt J, Sartor A, Thong-Vanh C, Valat-Rigot AS, Winer N, Lelong N, Khoshnood B; Prenatal MALFPULM Study Group. Prenatal natural history of congenital pulmonary malformations: MALFPULM population-based cohort study. Ultrasound Obstet Gynecol. 2019 Sep;54(3):381-388. doi: 10.1002/uog.20130. PMID 30264541
- [Derived] Weber M, Monier I, Rahshenas M, Salomon LJ, Sananes N, Castaigne V, Houfflin-Debarge V, Jouannic JM, Massardier J, Tsatsaris V, Khoshnood B, Lelong N; MALFPULM study group; Delacourt C, Benachi A. Fetal Therapy for Congenital Pulmonary Malformations: A Prospective Population-Based National Cohort Study. Prenat Diagn. 2024 Nov;44(12):1536-1547. doi: 10.1002/pd.6646. Epub 2024 Aug 13. PMID 39138024